CLINICAL TRIAL: NCT02810028
Title: Acceptance and Commitment Therapy for Muscle Disease
Acronym: ACTMuS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Barts & The London NHS Trust (Other); Muscular Dystrophy Association (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB-PG-061331085
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Muscle Diseases
Keywords: Limb girdle muscular dystrophy; Becker's muscular dystrophy; Facioscapulohumeral muscular dystrophy; Inclusion-body myositis; Acceptance and Commitment Therapy; ACT
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Muscular Dystrophy, Duchenne; Muscular Dystrophy, Facioscapulohumeral; Myositis, Inclusion Body | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT + Standard Medical Care (SMC) (Experimental): This consists of 4 self-guided psycho-education modules supported by weekly telephone contact with a health professional trained in Acceptance and Commitment Therapy (ACT). Standard medical care will be provided as usual.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Standard Medical Care (SMC) (No Intervention): All participants will receive SMC. As such, they will receive all the treatment and support they would otherwise receive outside of a research trial including a personalised assessment from the physiotherapist.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and Commitment Therapy (ACT) is a form of cognitive behavioural therapy focused explicitly on promoting psychological flexibility. An ACT programme suits the aims of the study because it targets avoidance of distress, promotes acceptance of illness through motivating meaningful activity outside of illness, improves the processes that underlie beliefs rather than by directly challenging beliefs, thus reducing possible trivialisation of the understandable distress caused by living with MD.
  Arms: ACT + Standard Medical Care (SMC)

SUMMARY:
In adults, muscle diseases are usually chronic long-term conditions that do not have a definitive cure. Supportive care has been shown to reduce complications from muscle disease and improved survival in some cases. However, there has been limited research to evaluate interventions that may improve quality of life (QoL) with this patient group. The QoL of those with MD is not just affected by the severity of their MD but also a variety of psychological variables. Based upon the knowledge of these psychological variables the investigators feel that a particular type of psychological intervention known as "acceptance and commitment therapy" (ACT) could potentially improve QoL in those with MD. The investigators therefore propose to test whether ACT does in fact improve QoL in those with MD by randomising 154 patients to receive either standard medical care plus a guided self-help ACT programme, or standard medical care only.

DETAILED DESCRIPTION:
Previous research has shown that while QoL is determined by the severity of the MD, this does not explain all aspects of the reduced QoL of those with MD. Previous research suggested that a cognitive behavioural approach using Acceptance and Commitment Therapy (ACT) would best suit those with MD. A pilot study of this approach in seven participants with MD was promising, and has led to this definitive trial of ACT. The aim of this study is to determine the efficacy of an ACT intervention to improve the QoL of individuals with MD.

Patients with one of the following muscle diseases will be recruited: limb girdle muscular dystrophy, dystrophinopathies resulting in a Becker' muscular dystrophy phenotype, facioscapulohumeral muscular dystrophy and inclusion body myositis. Patients will be recruited primarily through muscle clinics at King's College Hospital (KCH) and The Royal London Hospital (RLH) but also via Muscular Dystrophy UK (MDUK) and UK registries of patients with these muscle diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with one of four specific muscle diseases on the basis of diagnostic criteria:

   1. Limb girdle muscular dystrophy; symptomatic limb girdle muscular dystrophy genetically or pathologically proven
   2. Dystrophinopathies resulting in a Becker' muscular dystrophy phenotype (excluding Duchenne muscular dystrophy) with pathology or genetic diagnosis
   3. Facioscapulohumeral muscular dystrophy diagnosed clinically with specific genetic abnormality in the subject or their family
   4. Inclusion body myositis clinic-pathologically defined, clinically defined or probable IBM based on ENMC research diagnostic criteria 2013 (submitted)
2. duration of muscle disease greater than six months
3. over the age of 18 years
4. access to the internet and a computer on which they can receive the intervention materials
5. HADS scores > 8 for depression or >8 for anxiety

Exclusion Criteria:

1. Major active co-morbidities unrelated to muscle disease such as arthritis, respiratory disease, cardiovascular disease
2. Unstable complications of muscle disease including:

   1. neuromuscular respiratory weakness
   2. cardiomyopathy
3. Cognitive impairment that prevents comprehension of the questionnaires; assessed using the Montreal Cognitive Assessment
4. Unable to read English questionnaires
5. Major diagnosed active mental health co-morbidities e.g. psychosis, major depression, obsessive compulsive disorder, active suicide risk
6. Current or recent participation in other treatment intervention studies (< 4 weeks after completion)
7. Currently receiving psychological support or psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-07; Primary Completion 2018-04 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Individualised Neuromuscular Quality of Life Questionnaire (INQoL) - Life areas | 9 weeks post randomisation
  Measures impact of MD on life areas: activities, independence, social functioning, emotional functioning and body image.

SECONDARY OUTCOMES:
Individualised Neuromuscular Quality of Life Questionnaire (INQoL) - Symptom impact domains | 9 weeks post randomisation
  Measures the impact of key muscle disease symptoms: weakness, fatigue and pain.
Work and Social Adjustment Scale (WSAS) | 9 weeks post randomisation
  Assesses how much symptoms interfere with participation in life i.e. work, home management, social, private and relationships.
Hospital Anxiety and Depression Scale (HADS) | 9 weeks post randomisation
  Measures mood.
Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) | 9 weeks post randomisation
  Measures functional impairment.
Acceptance and Action Questionnaire (AAQ-II) | 9 weeks post randomisation
  Measures psychological flexibility.
Mindfulness Attention Awareness Scale (MAAS) | 9 weeks post randomisation
  Measures dispositional open awareness of and attention to the present moment.
Committed Action Scale (CAS) | 9 weeks post randomisation
  Measures commitment towards goals.
IBM Functional Rating Scale | 9 weeks post randomisation
  Assesses function in people with Inclusion Body Myositis.
Patient Global Impression of Change scale (PGIC) | 9 weeks post randomisation
  Assesses patient's own impression of change during the course of the study.
Patient rating of treatment satisfaction | 9 weeks post randomisation
  Measures patient's satisfaction with the treatment they have received.

OTHER OUTCOMES:
6-minute timed walk test | Baseline only
  Measures mobility.
Adult Ambulatory Neuromuscular Assessment (AANA) | Baseline only
  An adult version of the North Star Ambulatory Assessment that measures motor function.
Manual Muscle Strength Testing (MMST) | Baseline only
  Measures muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rose, Principal Investigator — King's College Hospital NHS Trust; Trudie Chalder, Principal Investigator — King's College London; Lance McCracken, Principal Investigator — King's College London; Christopher Graham, Principal Investigator — University of Leeds; Sam Norton, Principal Investigator — King's College London; Aleksandar Radunovic, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- King's College Hospital; The Royal London Hospital; University Hospital Southampton; King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham CD, Gouick J, Krahe C, Gillanders D. A systematic review of the use of Acceptance and Commitment Therapy (ACT) in chronic disease and long-term conditions. Clin Psychol Rev. 2016 Jun;46:46-58. doi: 10.1016/j.cpr.2016.04.009. Epub 2016 Apr 20. PMID 27176925
- [Background] Graham CD, Gouick J, Ferreira N, Gillanders D. The influence of psychological flexibility on life satisfaction and mood in muscle disorders. Rehabil Psychol. 2016 May;61(2):210-7. doi: 10.1037/rep0000092. PMID 27196863
- [Background] Graham CD, Simmons Z, Stuart SR, Rose MR. The potential of psychological interventions to improve quality of life and mood in muscle disorders. Muscle Nerve. 2015 Jul;52(1):131-6. doi: 10.1002/mus.24487. Epub 2015 May 28. PMID 25297932
- [Background] Rose MR, Sadjadi R, Weinman J, Akhtar T, Pandya S, Kissel JT, Jackson CE; Muscle Study Group. Role of disease severity, illness perceptions, and mood on quality of life in muscle disease. Muscle Nerve. 2012 Sep;46(3):351-9. doi: 10.1002/mus.23320. PMID 22907225
- [Derived] Rose M, Graham CD, O'Connell N, Vari C, Edwards V, Taylor E, McCracken LM, Radunovic A, Rakowicz W, Norton S, Chalder T. A randomised controlled trial of acceptance and commitment therapy for improving quality of life in people with muscle diseases. Psychol Med. 2023 Jun;53(8):3511-3524. doi: 10.1017/S0033291722000083. Epub 2022 Feb 23. PMID 35192788
- [Derived] Rose MR, Norton S, Vari C, Edwards V, McCracken L, Graham CD, Radunovic A, Chalder T. Acceptance and Commitment Therapy for Muscle Disease (ACTMus): protocol for a two-arm randomised controlled trial of a brief guided self-help ACT programme for improving quality of life in people with muscle diseases. BMJ Open. 2018 Oct 3;8(10):e022083. doi: 10.1136/bmjopen-2018-022083. PMID 30287669